CLINICAL TRIAL: NCT02822690
Title: Research Into the Quality of the Dying Phase in Hospitals in the Province of Groningen
Brief Title: Research Into the Quality of the Dying Phase
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 2016pz/1
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cessation of Life
Keywords: palliative care; Quality of dying
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- University Medical Center Groningen: all patients that died on one of the wards with the exception of children; on several wards the Hospice care will be introduced as an intervention
  Interventions: Other: Hospice care at UMCG
- Martini Ziekenhuis: all patients that died on one of the wards with the exception of children
- Ommelander ZorgGroep: all patients that died on one of the wards with the exception of children

INTERVENTIONS:
Other: Hospice care at UMCG — introduction of hospice care facilities on the wards at the UMCG
  Groups: University Medical Center Groningen

SUMMARY:
The aim of this study is to get insight in the quality of life at the end of life and quality of dying for patients died at the hospital in the department Groningen (the Netherlands).

The primary endpoint is the quality of life at the end of life and the secondary endpoint is the quality of dying. Both according a numerical rating scale.

An explorative analysis will be done for differences for the hospitals in Groningen, effect of using the Liverpool care Pathway for the dying, effect of using consultation by the palliative consultation team, effect of using the Hospice@UMCG intervention, correlation with the quality of life at the end of life and quality of dying according to nurses and doctors.

DETAILED DESCRIPTION:
Three hospitals in the department Groningen (the Netherlands) will participate in this study. When a patient died in one of these hospitals (except the emergency department, child ward and intensive care unit) the bereaved relatives will get an information letter. After about 12 weeks a questionnaire will be sent to the bereaved relative. This questionnaire is developed to evaluate the end of life care at the hospital.

Shortly after the patient died at the hospital, also the nurse and doctor of this patient are requested to fill out a questionnaire.

The questionnaire for the bereaved relatives consists of items, divided in groups: a general part, followed by questions of the last days of life, existing symptoms (physical, psychological, existential and social), the care and treatment and the loss.

The questionnaire for the nurses exists of similar items. Special attention for recognizing the impending dying and problems, care and therapy at the end of life.

In all questionnaires there are also 2 main questions: What is your opinion of the quality of life during the last days of life and What is your opinion of the quality of dying.

In the three hospitals the end of life care is managed at somehow different ways: the use of the Liverpool care Pathway of the dying, the hospice@UMCG intervention and consultation by the palliative team of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients dying in the hospital

Exclusion Criteria:

* patients dying at the child ward, emergency dept. and intensive care dept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients dying in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-10; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No